CLINICAL TRIAL: NCT06217250
Title: Hot EMR vs Underwater Cold EMR for Large Colonic Adenomas (>20 mm): the "CO.W.L." Prospective Randomized Trial
Brief Title: Hot EMR vs Underwater Cold EMR for Large Colonic Adenomas
Acronym: COWL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COWL
Record Dates: First submitted 2023-11-09; First posted 2024-01-22 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2023-11

CONDITIONS: Colonic Neoplasms; Colonic Adenoma; Colonic Lesion
MeSH Terms: conditions — Colonic Neoplasms | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional EMR (Active Comparator): Conventional EMR with thermal ablation of resection margins: initial submucosal injection of saline and methylene blue and subsequent piecemeal resection with 10- or 15-mm diathermic snare with subsequent thermal ablation of resection margins with snare tip soft coagulation.
  Interventions: Procedure: Traditional EMR
- Underwater Cold EMR (Experimental): Underwater Cold EMR (CS-EMR): after filling the lumen with water, initial submucosal injection of saline and methylene blue and subsequent piece-meal resection carried out with dedicated cold snare.
  Interventions: Procedure: the cold snare ("CO"), underwater technique ("W"), and the use of submucosal lift ("L") in both study arms

INTERVENTIONS:
Procedure: Traditional EMR — Conventional EMR with thermal ablation of resection margins: initial submucosal injection of saline and methylene blue and subsequent piecemeal resection with 10- or 15-mm diathermic snare with subsequent thermal ablation of resection margins with snare tip soft coagulation.Nevertheless, this technique is associated with the emergence of serious adverse events (SAEs), including delayed bleeding (PPB), electrocautery-induced post-polipectomy syndrome (PPS), and perforation(4).
  Other Names: Endoscopic Mucosal Resection
  Arms: Conventional EMR
Procedure: the cold snare ("CO"), underwater technique ("W"), and the use of submucosal lift ("L") in both study arms — The "cold-EMR" technique, as opposed to the conventional approach, employs a specialized snare that enables tissue transection without the need for electrical current, particularly in appropriately selected lesions. This approach yields the same efficacy outcome as the conventional procedure but offers the advantage of reducing the risks associated with polypectomy, which are often secondary to the use of diathermic current. Subsequently, the lesion fragments are retrieved for histological examination. Furthermore, the use of underwater setting, as demonstrated for hot EMR, could improve the effectiveness of cold-EMR.
  Arms: Underwater Cold EMR

SUMMARY:
This randomized, multi-center trial aims to evaluate the advantages of underwater cold endoscopic mucosal resection technique (CS-EMR) in comparison to the conventional endoscopic mucosal resection technique (EMR) for laterally spreading colorectal lesions exceeding 20 mm in size. More precisely, our hypothesis posits that underwater cold EMR is non-inferior to conventional EMR in terms of recurrence rates, resection completeness and safety.

DETAILED DESCRIPTION:
Endoscopic mucosal resection stands as one of the most commonly employed techniques for the removal of gastrointestinal lesions, particularly within the colon. "Piece-meal" endoscopic mucosal resection is the preferred approach for large colonic polyps without signs of deep infiltration. This method consists of the removal of lesions in multiple fragments.

The conventional procedure starts with the initial submucosal infiltration of the submucosal layer using a physiological solution and methylene blue, forming a cushion that facilitates tissue transection with the assistance of a diathermic snare. The goal is to remove the lesions in larger fragments whenever possible.

In contrast, the "cold" procedure, employs a specialized snare that enables tissue transection without the need for electrical current. This approach yields the same outcome as the conventional procedure but offers the advantage of reducing the risks associated with the use of diathermic current. Subsequently, the lesion fragments are retrieved for histological examination.

ELIGIBILITY:
Inclusion criteria:

* all patients ≥ 18 years of age undergoing colonoscopy for any indication (screening, anaemia, surveillance)
* patients who were able to give informed written consent.

Exclusion criteria:

* lesions suspicious for submucosal invasion (e.g. Kudo V or Paris 0-IIa-IIc with nongranular surface).
* lesions with large (>10 mm) Paris 0-Is component that could compromise the nodular en-bloc resection and increase risk of submucosal invasion.
* suspected sessile serrated adenomas (SSAs) according to traditional features such as adherent surface mucus, cloud-like surface, interruption of mucosal vessels, Kudo II-o pit pattern.
* pedunculated polyps
* active/quiescent colitis
* patients with other lesions resected by hot snare during the same procedure.
* rectal lesions
* residual or recurrent adenoma after endoscopic mucosal resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2024-04-15 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Success rate of resection defined as absence of residual/recurrence in SC1 and/or SC2 | at 6 and/or 12 months

SECONDARY OUTCOMES:
technical success | 2 years
  defined by the complete resection of polyp
Rate of intraprocedural adverse events such as bleeding or perforation | 2 years
  Defined as any procedure-related complication that compromises the completeness of the procedure and/or results in unplanned hospitalization of the patient
Rate of delayed bleeding of the patient | 2 years
Rate of post-polipectomy syndrome | 2 years
Rate of delayed perforation | 2 years
Avarage time of procedure and polyp resection time | 2 years

REFERENCES:
- [Background] Nishihara R, Wu K, Lochhead P, Morikawa T, Liao X, Qian ZR, Inamura K, Kim SA, Kuchiba A, Yamauchi M, Imamura Y, Willett WC, Rosner BA, Fuchs CS, Giovannucci E, Ogino S, Chan AT. Long-term colorectal-cancer incidence and mortality after lower endoscopy. N Engl J Med. 2013 Sep 19;369(12):1095-105. doi: 10.1056/NEJMoa1301969. PMID 24047059
- [Background] Ferlitsch M, Moss A, Hassan C, Bhandari P, Dumonceau JM, Paspatis G, Jover R, Langner C, Bronzwaer M, Nalankilli K, Fockens P, Hazzan R, Gralnek IM, Gschwantler M, Waldmann E, Jeschek P, Penz D, Heresbach D, Moons L, Lemmers A, Paraskeva K, Pohl J, Ponchon T, Regula J, Repici A, Rutter MD, Burgess NG, Bourke MJ. Colorectal polypectomy and endoscopic mucosal resection (EMR): European Society of Gastrointestinal Endoscopy (ESGE) Clinical Guideline. Endoscopy. 2017 Mar;49(3):270-297. doi: 10.1055/s-0043-102569. Epub 2017 Feb 17. PMID 28212588
- [Background] Sidhu M, Shahidi N, Gupta S, Desomer L, Vosko S, Arnout van Hattem W, Hourigan LF, Lee EYT, Moss A, Raftopoulos S, Heitman SJ, Williams SJ, Zanati S, Tate DJ, Burgess N, Bourke MJ. Outcomes of Thermal Ablation of the Mucosal Defect Margin After Endoscopic Mucosal Resection: A Prospective, International, Multicenter Trial of 1000 Large Nonpedunculated Colorectal Polyps. Gastroenterology. 2021 Jul;161(1):163-170.e3. doi: 10.1053/j.gastro.2021.03.044. Epub 2021 Mar 31. PMID 33798525
- [Background] Russo P, Barbeiro S, Awadie H, Libanio D, Dinis-Ribeiro M, Bourke M. Management of colorectal laterally spreading tumors: a systematic review and meta-analysis. Endosc Int Open. 2019 Feb;7(2):E239-E259. doi: 10.1055/a-0732-487. Epub 2019 Jan 30. PMID 30705959
- [Background] Thoguluva Chandrasekar V, Aziz M, Patel HK, Sidhu N, Duvvuri A, Dasari C, Kennedy KF, Ashwath A, Spadaccini M, Desai M, Jegadeesan R, Sathyamurthy A, Vennalaganti P, Kohli D, Hassan C, Pellise M, Repici A, Sharma P, Bourke MJ. Efficacy and Safety of Endoscopic Resection of Sessile Serrated Polyps 10 mm or Larger: A Systematic Review and Meta-Analysis. Clin Gastroenterol Hepatol. 2020 Oct;18(11):2448-2455.e3. doi: 10.1016/j.cgh.2019.11.041. Epub 2019 Nov 29. PMID 31786330
- [Background] Spadaccini M, Alfarone L, Facciorusso A, Gkolfakis P, Thoguluva Chandrasekar V, Fugazza A, Colombo M, Capogreco A, Massimi D, Carrara S, Alkandari A, Bhandari P, Maselli R, Hassan C, Repici A. Cold-snare endoscopic resection of non-ampullary duodenal adenomas: Systematic review and pooled-analysis. Dig Liver Dis. 2024 Apr;56(4):656-662. doi: 10.1016/j.dld.2023.09.013. Epub 2023 Sep 28. PMID 37777353
- [Background] Ito A, Suga T, Ota H, Tateiwa N, Matsumoto A, Tanaka E. Resection depth and layer of cold snare polypectomy versus endoscopic mucosal resection. J Gastroenterol. 2018 Nov;53(11):1171-1178. doi: 10.1007/s00535-018-1446-2. Epub 2018 Mar 7. PMID 29516270
- [Background] Suresh S, Zhang J, Ahmed A, Abu Ghanimeh M, Elbanna A, Kaur R, Isseh M, Watson A, Dang DT, Chathadi KV, Pompa R, Singla S, Piraka C, Zuchelli T. Risk factors associated with adenoma recurrence following cold snare endoscopic mucosal resection of polyps >/= 20 mm: a retrospective chart review. Endosc Int Open. 2021 Jun;9(6):E867-E873. doi: 10.1055/a-1399-8398. Epub 2021 May 27. PMID 34079869
- [Background] Maruoka D, Kishimoto T, Matsumura T, Arai M, Akizue N, Ishikawa K, Ohta Y, Kasamatsu S, Taida T, Ishigami H, Okimoto K, Saito K, Nakagawa T, Kato N. Underwater cold snare polypectomy for colorectal adenomas. Dig Endosc. 2019 Nov;31(6):662-671. doi: 10.1111/den.13427. Epub 2019 May 27. PMID 31038769
- [Background] Forbes N, Gupta S, Frehlich L, Meng ZW, Ruan Y, Montori S, Chebaa BR, Dunbar KB, Heitman SJ, Feagins LA, Albeniz E, Pohl H, Bourke MJ. Clip closure to prevent adverse events after EMR of proximal large nonpedunculated colorectal polyps: meta-analysis of individual patient data from randomized controlled trials. Gastrointest Endosc. 2022 Nov;96(5):721-731.e2. doi: 10.1016/j.gie.2022.05.020. Epub 2022 Jun 3. PMID 35667388
- [Background] Rotermund C, Djinbachian R, Taghiakbari M, Enderle MD, Eickhoff A, von Renteln D. Recurrence rates after endoscopic resection of large colorectal polyps: A systematic review and meta-analysis. World J Gastroenterol. 2022 Aug 7;28(29):4007-4018. doi: 10.3748/wjg.v28.i29.4007. PMID 36157546
- [Background] Rex DK, Anderson JC, Pohl H, Lahr RE, Judd S, Antaki F, Lilley K, Castelluccio PF, Vemulapalli KC. Cold versus hot snare resection with or without submucosal injection of 6- to 15-mm colorectal polyps: a randomized controlled trial. Gastrointest Endosc. 2022 Aug;96(2):330-338. doi: 10.1016/j.gie.2022.03.006. Epub 2022 Mar 12. PMID 35288147